CLINICAL TRIAL: NCT00296699
Title: A Pilot Study Assessing Duloxetine's Efficacy in Atypical Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Jonathon W. Stewart, New York State Psychiatric Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB4943
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Atypical Depression
Keywords: Atypical Depression; Major Depressive Disorder; Dysthymic Disorder; Atypical Features; Duloxetine
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine — Day 1-7: 20 mg/d; day 8-24: 30 mg/d; day 15-28: 60 mg/d; day 29-56: 120 mg/d.
  * dose raises will occur only if pt. is tolerating the previous dose and not remitting.; dose may be lowered or increased in 30 mg increments if pt. has difficulty tolerating.
  Other Names: Cymbalta

SUMMARY:
This is a Pilot Study to get a first indication whether Duloxetine may be effective for depressed patients with Atypical Features.

DETAILED DESCRIPTION:
This Open Pilot Study will assess whether Duloxetine is effective for patients with Atypical Features. 20 patients having Major Depressive Disorder with Atypical Features or Dysthymic Disorder will receive Duloxetine in open fashion for 8 weeks. Dose will begin with 20 mg/d and increase to PDR maximal dose of 120 mg/d, if tolerated.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV Major Depression or Dysthymia with Atypical Features
* Age 18-65
* Physically healthy
* HAMD(24) > 14

Exclusion Criteria:

* Prior experience with Duloxetine
* History of Psychosis or Bipolar Disorder, Borderline Personality Disorder
* Unstable medical disorder; any history of Epilepsy
* Currently taking medication that can interact with Duloxetine
* Current (past six months) Substance Use Disorder (illicit drugs and/or alcohol)
* Serious suicidal ideation judged at least somewhat likely to be acted upon or require hospitalization
* Current (past two weeks) use of psychoactive medication (four weeks for Fluoxetine)
* Pregnancy
* Currently breast feeding
* Fecund women failing to use acceptable birth control
* Refractory Depression (defined as failure to respond to one or more adequate trials of marketed antidepressants [i.e., >=2/3 PDR maximum dose for at least 4 weeks] during current episode)
* Serious suicidal ideation, recent (past six months) suicidal activity, any life-time history of serious suicide attempt (e.g., admitted to ICU, any duration of coma)
* Currently taking medication deemed effective

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-03; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale (HAM-D) | 10 weeks

SECONDARY OUTCOMES:
Atypical Depression Diagnostic Scale (ADDS) | 10 weeks
Beck Depression Inventory (BDI) | 10 weeks
Clinical Global Impression (CGI) | 10 weeks
Patient Global Impression (PGI) | 10 weeks
Inventory of Depressive Symptoms(IDS) | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W. Stewart, M.D., Principal Investigator — New York State Psychiatric Institute - Columbia University Department of Psychiatry
Locations (1):
- Depression Evaluation Service - New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- See also: Depression Evaluation Service - official website — http://www.depression-nyc.org
- See also: New York State Psychiatric Institute - official website — http://www.nyspi.org